CLINICAL TRIAL: NCT05530889
Title: Evaluating Quality of Life Benefits of ACUVUE® Theravision® With Ketotifen in Subjects With Ocular Allergies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to changes in business priorities, CR-6494 has been withdrawn.
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-6494
Record Dates: First submitted 2022-08-29; First posted 2022-09-07 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Ocular Physiology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL (Experimental): Eligible subjects who suffer from ocular allergies and who wear contact lenses will be randomized into the wear sequence (TEST/CONTROL) to wear the study lenses during each dispensing period (12-16 days).
  Interventions: Device: TEST Lens; Device: CONTROL Lens
- CONTROL/TEST (Experimental): Eligible subjects who suffer from ocular allergies and who wear contact lenses will be randomized into the wear sequence (CONTROL/TEST) to wear the study lenses during each dispensing period (12-16 days).
  Interventions: Device: TEST Lens; Device: CONTROL Lens

INTERVENTIONS:
Device: TEST Lens — ACUVUE® Theravision® with Ketotifen
Device: CONTROL Lens — 1-DAY ACUVUE® MOIST.

SUMMARY:
This will be a prospective, randomized, bilateral eye, crossover, non-masked single site pilot study to compare the severity of symptoms of itching between test and control lens after two weeks of wear.

ELIGIBILITY:
Inclusion Criteria:

Potential participants must satisfy all of the following criteria to be enrolled in the study

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be at least 18 years of age at the time of screening.
4. By self-report, habitually wear soft, daily, spherical contact lenses in both eyes. Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 5 days per week during the last 4 weeks.
5. Willing to wear study lenses for at least 5 days per week and 6 hours per day.
6. Possess a wearable pair of spectacles that provide correction for distance vision and agree to wear them on the day of the dispense visit (V2).
7. Must agree and be willing to not wear their habitual contact lenses on the day of the lens dispense visit (V2)
8. Report symptoms of allergy, including itchy eyes.
9. Oral medication and/or eye drops to treat allergy symptoms must have been used for at least 2 weeks, for a minimum of 3 times per week, prior to the screening visit.
10. Must be willing to cease use of habitual eye drops to relieve allergy symptoms during the ACUVUE® Theravision® with Ketotifen wear period.
11. The spherical equivalent of the participant's vertex corrected distance refraction must be between -0.50 and -7.00 DS (inclusive) in each eye.
12. The magnitude of the cylindrical component of the participant's vertex-corrected distance refraction must be no more than -1.00 DC (inclusive) in each eye.
13. Must achieve best corrected visual acuity (BCVA) of at least +0.20 logMAR in each eye.

Exclusion Criteria:

Potential participants who meet any of the following criteria will be excluded from participating in the study:

1. Be currently using any ocular medications, with the exception of eye drops for the treatment of their allergy symptoms.
2. Take any medications for which a stable regimen has not been achieved (i.e. have started a new medication or changed dosage of an existing medication within the last four weeks).
3. Have a known hypersensitivity or allergic reaction to ketotifen or sodium fluorescein.
4. Have participated in a contact lens or lens care product clinical trial within 14 days prior to study enrollment.
5. Be an employee (e.g., Investigator, Coordinator, Technician) of the Centre for Ocular Research & Education listed on the study Delegation Log or immediate family member of these employees (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse).
6. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).
7. Be currently using bifocal, multifocal or monovision contact lenses, or wear lenses in an extended wear modality (sleep in lenses)
8. Have any active ocular infection of any type.
9. Have clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
10. Have clinically significant (grade 3 or 4) papillary conjunctivitis or bulbar injection which might interfere with contact lens wear and that are unlikely to be related to their ocular allergy (at the investigator's discretion).
11. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-05-13 (Estimated); Study Completion 2024-05-13 (Estimated)

PRIMARY OUTCOMES:
Subjective rating of itchiness | up to 2-week follow-up
  The severity of symptoms of itching will be compared (0-4 itching scale with 0.5 steps) between the test and control lens after 2 weeks of wear.

SECONDARY OUTCOMES:
Subjective rating of comfort | up to 2-week follow-up
  Subjective ratings of comfort will be assessed on a 0 to 100 scale after each 2-week wear period.
Subjective rating of dryness | up to 2-week follow-up
  Subjective ratings of dryness will be assessed on a 0 to 100 scale after each 2-week wear period.
Subjective rating of vision | up to 2-week follow-up
  Subjective ratings of vision will be assessed on a 0 to 100 scale after each 2-week wear period.
Subjective rating of handling | up to 2-week follow-up
  Subjective ratings of handling will be assessed on a 0 to 100 scale after each 2-week wear period.
CLDEQ-8 Questionnaire | up to 2-week follow-up
  CLDEQ-8 is a dry eye questionnaire that asks the participant to reflect and rate their symptoms of eye discomfort and dryness over the past two weeks. A higher composite score indicates more severe dryness and the range is 0-37.
Comfortable and total CL wear time | up to 2-week follow-up
  Total wearing time and total comfortable wearing time will be recorded after each 2-week wear period.
Subject Preference Questionnaire | at the 2-week follow-up
  The subject will select their preferred study lens, test lens or control lens.
MiniRQLQ Questionnaire | up to 2-week follow-up
  The MiniRQLQ is a validated questionnaire that focuses on the impact of allergies on quality of life (QoL). It includes 14 questionnaire items in five sections (activities, practical problems, nasal symptoms, ocular symptoms, general symptoms) that address how allergies impacted QoL during the previous week, by asking the user to rate how troubling each item in the questionnaire was perceived.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu